CLINICAL TRIAL: NCT02655029
Title: Prospective, Non-interventional Study for the Recording of Adherence to Treatment With Perindopril/Indapamide/Amlodipine Fixed Dose Combination, in a Greek Population With Hypertension
Brief Title: Study for the Recording of Adherence to Treatment With Perindopril/Indapamide/Amlodipine Fixed Dose Combination
Acronym: CONTROL-3
Status: Completed | Type: Observational
Sponsor: Servier Hellas Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: IC4-06593-021-GRC
Record Dates: First submitted 2016-01-05; First posted 2016-01-13 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Adherence to Medication Regime; Hypertensive Disease
MeSH Terms: conditions — Medication Adherence; Hypertension | interventions — Perindopril; Indapamide; Amlodipine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Perindopril/Indapamide/Amlodipine fixed dose combination — Dose selection is based on investigators management.
  Other Names: Triplixam

SUMMARY:
The main objective of this study is to record, in routine clinical practice, patients' adherence to treatment with Perindopril/Indapamide/Amlodipine fixed dose combination, during 4 months treatment.

DETAILED DESCRIPTION:
This is a non-interventional study aiming to record adherence to treatment with Perindopril/Indapamide/Amlodipine fixed dose combination. In parallel blood pressure levels will be recorded, as well as safety and tolerability of this fixed dose combination.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ambulatory patients >18 years old.
* Clinically diagnosed essential arterial hypertension.
* Under treatment with Perindoril/Indapamide/Amlodipine fixed dose combination.
* The patient has given his/her written consent after being informed, before his inclusion in the study.

Exclusion Criteria:

* Secondary arterial hypertension.
* Serious end stage diseases, severe neuropsychiatric diseases, cerebrovascular event with serious residual lesions, scheduled procedure or surgical operation or hospital admission.
* Pregnancy, lactation or intention to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greek patients with arterial hypertension who receive treatment with Perindopril/Indapamide/Amlodipine fixed dose combination.
Sampling Method: Probability Sample
Enrollment: 2285 (Actual)
Dates: Start 2015-11-25 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | Change of total score of compliance scale between baseline and 1st month and between 1st and 4th month of treatment
  Total score of Hill-Bone High Blood Pressure Compliance Scale will be recorded at each study visit

SECONDARY OUTCOMES:
Systolic Blood Pressure | All visits (baseline, 1st and 4th month of treatment)
Diastolic Blood Pressure | All visits (baseline, 1st and 4th month of treatment)
Adverse events recording leading to treatment discontinuation | 1st and 4th month of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Tsioufis, Professor, Principal Investigator — Ippokrateion General Hospital of Athens
Locations (1):
- Ippokratio University Hospital of Athens, Athens, Greece